CLINICAL TRIAL: NCT01273103
Title: An Open Label, Single Dose, Mass Balance Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C-GSK2248761 200 mg, Administered as an Oral Suspension to Healthy Adult Subjects
Brief Title: A Study to Investigate the Recovery, Excretion, and Pharmacokinetics of 14C-GSK2248761 Administered as an Oral Suspension to Healthy Adult Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: GSK2248761 development program is on clinical hold.
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 113393
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): [14C]- GSK2248761 200 mg
  Interventions: Drug: 200mg [14C]- GSK2248761

INTERVENTIONS:
Drug: 200mg [14C]- GSK2248761 — single oral suspension dose of [14C]- GSK2248761 200 mg

SUMMARY:
This study is a Phase I, open-label, single dose, mass balance study in a cohort of 6 healthy adult male subjects. The study will consist of: Screening evaluations, a treatment phase, and follow-up evaluations. In the treatment phase, after an overnight fast of at least 10 hours, each subject will receive a single oral suspension dose of GSK2248761 200mg containing [14C] - GSK2248761. Following dosing, serial whole blood, plasma, urine, and fecal samples will be collected. Subjects will be required to remain in the unit until the radiocarbon excreted falls to less than or equal to 1% of the administered dose for two consecutive 24-hour collections in both urine and feces, whichever occurs first. Safety will be assessed by vital signs, 12-lead electrocardiogram (ECG), clinical laboratory tests, AE monitoring, and physical examinations as indicated.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male subjects between 30 and 55 years of age.
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 84 days after the dose of study medication. Male subjects also must refrain from the donation of sperm during this time as well.
* Body weight greater than or equal to 50 kg and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Available to complete the study (minimum of 7 and a maximum of 11 night's confinement in the clinical research unit).
* A history of regular bowel movements (averaging one or more bowel movements per day).
* AST, ALT, alkaline phosphatase and bilirubin greater than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.

Exclusion Criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including antacids, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study
* Has a history or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Subjects who have received a total body radiation dose of greater than 5.0 mSv (upper limit of WHO category II) or exposure to significant radiation (e.g. serial x-ray or CT scans, barium meal etc) in the 12 months prior to this study. Any previous radiolabeled study drug must have been received more than 6 months prior to check-in. Also the total exposure from this current study and any previous studies must be within the recommended levels considered safe of 5 Rems whole body annual exposure, as per United States (US) Code of Federal Regulations (CFR) 21 CFR 361.1.
* Any condition that could interfere with the accurate assessment and recovery of radiocarbon [14C].
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 45-100 bpm. A single repeat is allowed to determine eligibility.
* An abnormal ECG as specified in the protocol (a single repeat is allowed for eligibility determination).

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Percent recovery of total radiocarbon in urine and feces | up to 10 days
Area under the concentration-time curve from time zero to last time of quantifiable concentration within a subject (AUC (0-t)) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
Area under the concentration-time curve from time zero extrapolated to infinite time (AUC (0-infinity)) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
Percentage of AUC(0-infinity) obtained by extrapolation (%AUCex) of total drug-related material (radiocarbon) in blood and plasma. | up to 10 days
Minimum observed concentration (Cmax) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
Time occurence of Cmax (tmax) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
Terminal phase rate constant (lambda z) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
Lag time before observation of drug concentrations in sampled matrix (tlag) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
Terminal phase half life (t1/2) of total drug-related material (radiocarbon) in blood and plasma | up to 10 days
AUC (0-t) of GSK2248761 in plasma | up to 10 days
AUC (0-infinity) of GSK2248761 in plasma | up to 10 days
%AUCex of GSK2248761 in plasma | up to 10 days
Cmax of GSK2248761 in plasma | up to 10 days
tmax of GSK2248761 in plasma | up to 10 days
Lambda z of GSK2248761 in plasma | up to 10 days
tlag of GSK2248761 in plasma | up to 10 days
Apparent clearance following oral dosing (CL/F) of GSK2248761 in plasma | up to 10 days
Apparent volume of distribution after oral administration (Vz/F) of GSK2248761 in plasma | up to 10 days
t1/2 of GSK2248761 in plasma | up to 10 days

SECONDARY OUTCOMES:
Safety and tolerability parameters including number of adverse events (AEs) | up to 25 days
Safety and tolerability parameters including change from baseline for vital signs (blood pressure and heart rate) | up to 25 days
Safety and tolerability parameters including change from baseline for electrocardiogram assessments (ECGs) | up to 25 days
Safety and tolerability parameters including change from baseline for clinical laboratory assessments | up to 25 days
Blood:plasma ratio of total drug-related material (radioactivity) | up to 10 days
Percent of total radiocarbon associated with red blood cells | up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Madison, Wisconsin, United States